CLINICAL TRIAL: NCT04855513
Title: Prevention of Pre-eclampsia Using Metformin: a Randomized Control Trial
Acronym: PREMET
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hamad Medical Corporation (Industry)
Collaborators: Sidra Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IRGC-04-JI-17-164
Record Dates: First submitted 2021-04-19; First posted 2021-04-22 (Actual); Last update posted 2022-03-29 (Actual); Status verified 2022-03

CONDITIONS: Preeclampsia; Preeclampsia Severe; High Risk Pregnancy; Eclampsia
Keywords: Metformin
MeSH Terms: conditions — Pre-Eclampsia; Eclampsia | interventions — Metformin

STUDY DESIGN:
Intervention Model Description: A randomized control trial into two groups using block randomization based on predefined criteria
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- standard care (No Intervention): The control group will receive standard care treatment including aspirin according to ACOG guidelines. The control group estimated number of enrollment is 207 patients.
- Metformin (Experimental): The intervention group will be give metformin 500 mg orally three times daily in addition to standard of care. The estimated number to be enrolled are 207 patients.
  Interventions: Drug: Metformin

INTERVENTIONS:
Drug: Metformin — Metformin is a medication used for treatment of diabetes. In this study it will be used to explore is potential role in prevention of preeclampsia. The drug will start before 12 week of pregnancy and continue till delivery
  Other Names: Glucophage
  Arms: Metformin

SUMMARY:
This is an open label, randomized control trial (RCT) in which high risk for pre-eclampsia pregnant subjects will be randomly assigned to either an intervention group (metformin 1 gm twice daily plus aspirin 100 mg per day and standard of care) versus control group (aspirin 100 mg per day and standard of care) that will be administered between 11 to 13 weeks of gestation until delivery . Only women at high risk of pre-eclampsia as defined by the ACOG practice bulletin will be included (see inclusion criteria). Patient assignment will not be blinded as control group will not be given a placebo; the data will be analyzed on an intention to treat basis. Enrolled subjects will be followed throughout pregnancy and up to 30 days post-delivery (as per hospital practice).

DETAILED DESCRIPTION:
Preeclampsia (PET) is one of the leading causes of maternal morbidity and mortality . Its pathophysiology is poorly understood. Consequently, there are no efficient preventive and treatment modality. PET is associated with significant perinatal morbidity and mortality including prolonged hospitalization and is a major contributor to a large proportion of iatrogenic preterm birth. Women who suffer from PET are at a greater risk of hypertensive and cardiovascular diseases in later life and more likely to suffer from premature death. Since the only treatment for PET is delivery, a logical approach to reducing the incidence and therefore consequences is prevention. For this to be effective those at risk have to be identified and any timely interventions introduced.

Amongst the risk factors are maternal age, obesity, medical disorders such as antiphospholipid syndrome, hypertensive disorders, renal diseases diabetes mellitus and previous PET. A history of PET increases the risk of recurrence 7 fold and this is compounded by GA at delivery for the affected pregnancy . Moreover, both chronic hypertension and pre-existing diabetes increase the risk of PET which is further enhanced by the degree of glycemic control. Interestingly maternal and paternal history of diabetes and hypertension have been associated with increased risk of PET. Additionally, maternal age > 40 years and pregnancy interval > 10 years increases the risk of PET by two to three folds respectively .A BMI > 35 increases the risk of PET by 4 folds in both multiparous and nulliparous women. Moreover, assisted reproduction techniques and multiple gestation have also been associated with increased risk of PET. A combination of diabetes and obesity, which has a high prevalence in Qatar, significantly increases the risk of PET. Despite these risk factors only a fraction of those with at high risk eventually develop PET as the current criteria for prediction is not specific.

Various measures to predict, prevent and treat pre-eclampsia have been investigated and tried by several groups/researchers. However, these have not been very successful, primarily because PET is a disease of theories with an unclear primary pathophysiology and thus no clear target for either these predictive tools or interventions. Evidence, however, does suggest that in patients at risk of developing PET there is inadequate trophoblastic invasion, placental hypo-perfusion, and endothelial cell activation . This the basis for the most widely noninvasive clinical tool of Doppler velocimetry of the uterine artery; but again, this has a poor sensitivity. An imbalance in pro-angiogenic factors such as vascular endothelial growth factor (VEGF) and placental growth factor (PIGF) (decreased) and antiangiogenic factors such as soluble FMSlike tyrosine kinase -1 (sFlt-1) (increased) has been implicated for the inadequate remodeling of spiral arteries (which is essential for the maintenance of a normal placental perfusion) in women who develop PET.

Vascular endothelial growth factor (VEGF) is an important signaling protein in health and diseases such as cancer, kidney diseases and PET . The VEGF family is composed of five members and three tyrosine kinase receptors. The signaling proteins are: VEGFA, VEGFB,VEGFC, VEGFD and placental growth factor (PlGF) (reviewed in (20)). The receptor tyrosine kinase consists of VEGFR1 (also known as Flt-1), VEGFR2 and VEGF3, with different binding capacity to VEGF proteins . A soluble Fms like tyrosine kinase-1 (sFlt-1) a truncated form of VEGFR1, has also been identified which lacks the VEGFR1 cytosolic domain. In addition to ligand binding, VEGFR has been shown to be activated through non-ligand binding and mechanical forces. VEGF proteins are upregulated under hypoxic conditions such as PET, growth factor signaling and by hormones such as estrogen .PET is characterized by a hypoxic environment, resulting in considerable changes in maternal leukocyte gene expression, altered expression of the VEGF signaling pathway and AMPactivated protein kinase (AMPK) and secretion of sFlt-1 into the maternal circulation.VEGF including PIGF has been identified as a crucial in the signaling pathway for angiogenesis and vasculogenesis during placental development .Indeed, deletion of a single VEGF allele in mice resulted in embryonic lethality due to immature angiogenesis. The invasion of maternal spiral arteries by cytotrophoblasts is vital for adequate oxygen and nutrient supply . This process is believed to be mediated by binding of VEGF and PIGF to Flt-1 . Further, fetal DNA variants at the Flt-1 region has been associated with PET and reported recently . However, the pathophysiology of PET is still unclear and understanding of its molecular mechanism is warranted. A decreased level of VEGF and PIGF free form has been observed that has been attributed to their blockade by the increased level of sFlt-1 in pre-eclamptic women . Indeed, the introduction of sFlt-1 to a pregnant rat led to hypertension and proteinuria similar to that seen in PET women . Furthermore, an altered ratio of serum PIGF/sFlt-1 has been found to be associated with PET diagnosis and disease severity . Indeed, there is now a drive to use this ratio in screening women at risk of PET but most of the data were generated in late pregnancy rather than in early pregnancy - a time when interventions have been shown to have maximum impact . It would seem from this greater understanding of the underlying physiological changes in women that develop PET that any interventions that have the potential to alter this milieu are more likely to be successful .Very recently a double-blind, placebo-controlled trial, that randomly assigned pregnant women without diabetes who had a body-mass index of more than 35 to receive metformin, at a dose of 3.0 g per day, or placebo (225 women in each group) from 12 to 18 weeks of gestation until delivery showed a significant reduction in the incidence of PET in those who received metformin . Since metformin is now frequently prescribed to obese type II diabetic women and gestational diabetics with poor glycemic control on diet, it is hypothesized in those at risk of PET, metformin will not only reduce the incidence of PET but will modify the PIGF/s-Flt-1 ratio in favor of normal pregnancies.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed pregnancy
* Gestational age < 12+0 weeks
* Live fetus at time of booking ultrasound scan (between 11+0 and 13+6 weeks of gestation)
* To be considered as high risk of preeclampsia

Exclusion Criteria:

* Age under 18 years
* Hyperemesis gravidarum
* Unable to sign the consent form
* Type 1 or 2 diabetes mellitus
* Early gestational diabetes
* Auto-immune disease
* Fetal abnormality identified at time of scanning (between 11+0 and 13+6 weeks of gestation)
* Bleeding disorder
* Peptic ulcer
* Hypersensitivity to aspirin or metformin
* Long use of NSAIDS before initiation of intervention
* Contraindication to metformin or aspirin and participation in another concurrent trial.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Because the study will be on pregnant women
Enrollment: 414 (Estimated)
Dates: Start 2022-03-24 (Estimated); Primary Completion 2023-04-24 (Estimated); Study Completion 2023-12-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of PET | Through study completion period (3 years)
  To compare the incidence of PET between the metformin group (intervention group) versus control group
Evaluating PIGF/sFlt-1 as a prognostic marker in PET in Qatar | Through study completion period (3 years)
  Comparing PIGF/sFlt-1 ratio in both groups before and after developing PET

SECONDARY OUTCOMES:
PIGF/sFlt-1 as a prognostic marker in PET patients | Through study completion period (3 years)
  Comparing PIGF/sFlt-1 ratio in PET patients who received metformin versus PET patient in the standard care group
Maternal outcomes | Through study completion period (3 years)
  Comparing gestational age at PET onset, gestation age at delivery and PET severity between study groups

CONTACTS AND LOCATIONS:
Overall Officials: Mahmoud Mohamed, MSc, Principal Investigator — Hamad Medical Corporation; Justin Konje, MD, PhD, Study Chair — Hamad Medical Corporation; Mohamed Bashir, MD, Study Director — Hamad Medical Corporation; Damien Chausabel, PhD, Study Director — Sidra Medicine; Bara Al Jarrah, BSE, Study Director — Hamad Medical Corporation
Locations (1):
- Women Wellness and Research Center, Doha, Qatar

REFERENCES:
- [Background] Bartsch E, Medcalf KE, Park AL, Ray JG; High Risk of Pre-eclampsia Identification Group. Clinical risk factors for pre-eclampsia determined in early pregnancy: systematic review and meta-analysis of large cohort studies. BMJ. 2016 Apr 19;353:i1753. doi: 10.1136/bmj.i1753. PMID 27094586
- [Background] Duckitt K, Harrington D. Risk factors for pre-eclampsia at antenatal booking: systematic review of controlled studies. BMJ. 2005 Mar 12;330(7491):565. doi: 10.1136/bmj.38380.674340.E0. Epub 2005 Mar 2. PMID 15743856
- [Background] Mostello D, Kallogjeri D, Tungsiripat R, Leet T. Recurrence of preeclampsia: effects of gestational age at delivery of the first pregnancy, body mass index, paternity, and interval between births. Am J Obstet Gynecol. 2008 Jul;199(1):55.e1-7. doi: 10.1016/j.ajog.2007.11.058. Epub 2008 Feb 15. PMID 18280450
- [Background] Chappell LC, Enye S, Seed P, Briley AL, Poston L, Shennan AH. Adverse perinatal outcomes and risk factors for preeclampsia in women with chronic hypertension: a prospective study. Hypertension. 2008 Apr;51(4):1002-9. doi: 10.1161/HYPERTENSIONAHA.107.107565. Epub 2008 Feb 7. PMID 18259010
- [Background] Sibai BM, Caritis S, Hauth J, Lindheimer M, VanDorsten JP, MacPherson C, Klebanoff M, Landon M, Miodovnik M, Paul R, Meis P, Dombrowski M, Thurnau G, Roberts J, McNellis D. Risks of preeclampsia and adverse neonatal outcomes among women with pregestational diabetes mellitus. National Institute of Child Health and Human Development Network of Maternal-Fetal Medicine Units. Am J Obstet Gynecol. 2000 Feb;182(2):364-9. doi: 10.1016/s0002-9378(00)70225-0. PMID 10694338
- [Background] Qiu C, Williams MA, Leisenring WM, Sorensen TK, Frederick IO, Dempsey JC, Luthy DA. Family history of hypertension and type 2 diabetes in relation to preeclampsia risk. Hypertension. 2003 Mar;41(3):408-13. doi: 10.1161/01.HYP.0000056996.25503.F5. Epub 2003 Feb 17. PMID 12623936
- [Background] Bianco A, Stone J, Lynch L, Lapinski R, Berkowitz G, Berkowitz RL. Pregnancy outcome at age 40 and older. Obstet Gynecol. 1996 Jun;87(6):917-22. doi: 10.1016/0029-7844(96)00045-2. PMID 8649698
- [Background] Skjaerven R, Wilcox AJ, Lie RT. The interval between pregnancies and the risk of preeclampsia. N Engl J Med. 2002 Jan 3;346(1):33-8. doi: 10.1056/NEJMoa011379. PMID 11778000
- [Background] Wang Z, Wang P, Liu H, He X, Zhang J, Yan H, Xu D, Wang B. Maternal adiposity as an independent risk factor for pre-eclampsia: a meta-analysis of prospective cohort studies. Obes Rev. 2013 Jun;14(6):508-21. doi: 10.1111/obr.12025. Epub 2013 Mar 26. PMID 23530552
- [Background] Skupski DW, Nelson S, Kowalik A, Polaneczky M, Smith-Levitin M, Hutson JM, Rosenwaks Z. Multiple gestations from in vitro fertilization: successful implantation alone is not associated with subsequent preeclampsia. Am J Obstet Gynecol. 1996 Oct;175(4 Pt 1):1029-32. doi: 10.1016/s0002-9378(96)80047-0. PMID 8885770
- [Background] Chaiworapongsa T, Chaemsaithong P, Korzeniewski SJ, Yeo L, Romero R. Pre-eclampsia part 2: prediction, prevention and management. Nat Rev Nephrol. 2014 Sep;10(9):531-40. doi: 10.1038/nrneph.2014.103. Epub 2014 Jul 8. PMID 25003612
- [Background] Walsh SW. What causes endothelial cell activation in preeclamptic women? Am J Pathol. 2006 Oct;169(4):1104-6. doi: 10.2353/ajpath.2006.060713. No abstract available. PMID 17003470
- [Background] Goldman-Wohl D, Yagel S. Regulation of trophoblast invasion: from normal implantation to pre-eclampsia. Mol Cell Endocrinol. 2002 Feb 22;187(1-2):233-8. doi: 10.1016/s0303-7207(01)00687-6. PMID 11988332
- [Background] Gathiram P, Moodley J. Pre-eclampsia: its pathogenesis and pathophysiolgy. Cardiovasc J Afr. 2016 Mar-Apr;27(2):71-8. doi: 10.5830/CVJA-2016-009. PMID 27213853
- [Background] Nagar T, Sharma D, Choudhary M, Khoiwal S, Nagar RP, Pandita A. The Role of Uterine and Umbilical Arterial Doppler in High-risk Pregnancy: A Prospective Observational Study from India. Clin Med Insights Reprod Health. 2015 Apr 15;9:1-5. doi: 10.4137/CMRH.S24048. eCollection 2015. PMID 25922590
- [Background] Bates DO. An unexpected tail of VEGF and PlGF in pre-eclampsia. Biochem Soc Trans. 2011 Dec;39(6):1576-82. doi: 10.1042/BST20110671. PMID 22103490
- [Background] Herraiz I, Simon E, Gomez-Arriaga PI, Martinez-Moratalla JM, Garcia-Burguillo A, Jimenez EA, Galindo A. Angiogenesis-Related Biomarkers (sFlt-1/PLGF) in the Prediction and Diagnosis of Placental Dysfunction: An Approach for Clinical Integration. Int J Mol Sci. 2015 Aug 13;16(8):19009-26. doi: 10.3390/ijms160819009. PMID 26287164
- [Background] Shibuya M. VEGF-VEGFR Signals in Health and Disease. Biomol Ther (Seoul). 2014 Jan;22(1):1-9. doi: 10.4062/biomolther.2013.113. PMID 24596615
- [Background] Simons M, Gordon E, Claesson-Welsh L. Mechanisms and regulation of endothelial VEGF receptor signalling. Nat Rev Mol Cell Biol. 2016 Oct;17(10):611-25. doi: 10.1038/nrm.2016.87. Epub 2016 Jul 27. PMID 27461391
- [Background] Shibuya M, Yamaguchi S, Yamane A, Ikeda T, Tojo A, Matsushime H, Sato M. Nucleotide sequence and expression of a novel human receptor-type tyrosine kinase gene (flt) closely related to the fms family. Oncogene. 1990 Apr;5(4):519-24. PMID 2158038
- [Background] Parker MW, Xu P, Li X, Vander Kooi CW. Structural basis for selective vascular endothelial growth factor-A (VEGF-A) binding to neuropilin-1. J Biol Chem. 2012 Mar 30;287(14):11082-9. doi: 10.1074/jbc.M111.331140. Epub 2012 Feb 7. PMID 22318724
- [Background] Jin ZG, Ueba H, Tanimoto T, Lungu AO, Frame MD, Berk BC. Ligand-independent activation of vascular endothelial growth factor receptor 2 by fluid shear stress regulates activation of endothelial nitric oxide synthase. Circ Res. 2003 Aug 22;93(4):354-63. doi: 10.1161/01.RES.0000089257.94002.96. Epub 2003 Jul 31. PMID 12893742
- [Background] Tzima E, Irani-Tehrani M, Kiosses WB, Dejana E, Schultz DA, Engelhardt B, Cao G, DeLisser H, Schwartz MA. A mechanosensory complex that mediates the endothelial cell response to fluid shear stress. Nature. 2005 Sep 15;437(7057):426-31. doi: 10.1038/nature03952. PMID 16163360
- [Background] Gu Y, Lewis DF, Wang Y. Placental productions and expressions of soluble endoglin, soluble fms-like tyrosine kinase receptor-1, and placental growth factor in normal and preeclamptic pregnancies. J Clin Endocrinol Metab. 2008 Jan;93(1):260-6. doi: 10.1210/jc.2007-1550. Epub 2007 Oct 23. PMID 17956952
- [Background] Li H, Gu B, Zhang Y, Lewis DF, Wang Y. Hypoxia-induced increase in soluble Flt-1 production correlates with enhanced oxidative stress in trophoblast cells from the human placenta. Placenta. 2005 Feb-Mar;26(2-3):210-7. doi: 10.1016/j.placenta.2004.05.004. PMID 15708122
- [Background] Kaufman MR, Brown TL. AMPK and Placental Progenitor Cells. Exp Suppl. 2016;107:73-79. doi: 10.1007/978-3-319-43589-3_4. PMID 27812977
- [Background] Koga K, Osuga Y, Yoshino O, Hirota Y, Ruimeng X, Hirata T, Takeda S, Yano T, Tsutsumi O, Taketani Y. Elevated serum soluble vascular endothelial growth factor receptor 1 (sVEGFR-1) levels in women with preeclampsia. J Clin Endocrinol Metab. 2003 May;88(5):2348-51. doi: 10.1210/jc.2002-021942. PMID 12727995
- [Background] Brownfoot FC, Hastie R, Hannan NJ, Cannon P, Tuohey L, Parry LJ, Senadheera S, Illanes SE, Kaitu'u-Lino TJ, Tong S. Metformin as a prevention and treatment for preeclampsia: effects on soluble fms-like tyrosine kinase 1 and soluble endoglin secretion and endothelial dysfunction. Am J Obstet Gynecol. 2016 Mar;214(3):356.e1-356.e15. doi: 10.1016/j.ajog.2015.12.019. Epub 2015 Dec 22. PMID 26721779
- [Background] Rajakumar A, Chu T, Handley DE, Bunce KD, Burke B, Hubel CA, Jeyabalan A, Peters DG. Maternal gene expression profiling during pregnancy and preeclampsia in human peripheral blood mononuclear cells. Placenta. 2011 Jan;32(1):70-8. doi: 10.1016/j.placenta.2010.10.004. Epub 2010 Nov 13. PMID 21075447
- [Background] Wang Y, Zhao S. Vascular Biology of the Placenta. San Rafael (CA): Morgan & Claypool Life Sciences; 2010. Available from http://www.ncbi.nlm.nih.gov/books/NBK53247/ PMID 21452443
- [Background] Achen MG, Gad JM, Stacker SA, Wilks AF. Placenta growth factor and vascular endothelial growth factor are co-expressed during early embryonic development. Growth Factors. 1997;15(1):69-80. doi: 10.3109/08977199709002113. PMID 9401819
- [Background] Carmeliet P, Moons L, Luttun A, Vincenti V, Compernolle V, De Mol M, Wu Y, Bono F, Devy L, Beck H, Scholz D, Acker T, DiPalma T, Dewerchin M, Noel A, Stalmans I, Barra A, Blacher S, VandenDriessche T, Ponten A, Eriksson U, Plate KH, Foidart JM, Schaper W, Charnock-Jones DS, Hicklin DJ, Herbert JM, Collen D, Persico MG. Synergism between vascular endothelial growth factor and placental growth factor contributes to angiogenesis and plasma extravasation in pathological conditions. Nat Med. 2001 May;7(5):575-83. doi: 10.1038/87904. PMID 11329059
- [Background] Carmeliet P, Ferreira V, Breier G, Pollefeyt S, Kieckens L, Gertsenstein M, Fahrig M, Vandenhoeck A, Harpal K, Eberhardt C, Declercq C, Pawling J, Moons L, Collen D, Risau W, Nagy A. Abnormal blood vessel development and lethality in embryos lacking a single VEGF allele. Nature. 1996 Apr 4;380(6573):435-9. doi: 10.1038/380435a0. PMID 8602241
- [Background] Ferrara N, Carver-Moore K, Chen H, Dowd M, Lu L, O'Shea KS, Powell-Braxton L, Hillan KJ, Moore MW. Heterozygous embryonic lethality induced by targeted inactivation of the VEGF gene. Nature. 1996 Apr 4;380(6573):439-42. doi: 10.1038/380439a0. PMID 8602242
- [Background] Luttun A, Carmeliet P. Soluble VEGF receptor Flt1: the elusive preeclampsia factor discovered? J Clin Invest. 2003 Mar;111(5):600-2. doi: 10.1172/JCI18015. No abstract available. PMID 12618513
- [Background] King BF. Ultrastructural differentiation of stromal and vascular components in early macaque placental villi. Am J Anat. 1987 Jan;178(1):30-44. doi: 10.1002/aja.1001780105. PMID 2435141
- [Background] Zhou Y, McMaster M, Woo K, Janatpour M, Perry J, Karpanen T, Alitalo K, Damsky C, Fisher SJ. Vascular endothelial growth factor ligands and receptors that regulate human cytotrophoblast survival are dysregulated in severe preeclampsia and hemolysis, elevated liver enzymes, and low platelets syndrome. Am J Pathol. 2002 Apr;160(4):1405-23. doi: 10.1016/S0002-9440(10)62567-9. PMID 11943725
- [Background] Levine RJ, Maynard SE, Qian C, Lim KH, England LJ, Yu KF, Schisterman EF, Thadhani R, Sachs BP, Epstein FH, Sibai BM, Sukhatme VP, Karumanchi SA. Circulating angiogenic factors and the risk of preeclampsia. N Engl J Med. 2004 Feb 12;350(7):672-83. doi: 10.1056/NEJMoa031884. Epub 2004 Feb 5. PMID 14764923
- [Background] Maynard SE, Min JY, Merchan J, Lim KH, Li J, Mondal S, Libermann TA, Morgan JP, Sellke FW, Stillman IE, Epstein FH, Sukhatme VP, Karumanchi SA. Excess placental soluble fms-like tyrosine kinase 1 (sFlt1) may contribute to endothelial dysfunction, hypertension, and proteinuria in preeclampsia. J Clin Invest. 2003 Mar;111(5):649-58. doi: 10.1172/JCI17189. PMID 12618519
- [Background] Yusuf AM, Kahane A, Ray JG. First and Second Trimester Serum sFlt-1/PlGF Ratio and Subsequent Preeclampsia: A Systematic Review. J Obstet Gynaecol Can. 2018 May;40(5):618-626. doi: 10.1016/j.jogc.2017.07.014. Epub 2017 Sep 15. PMID 28927814
- [Background] Chang YS, Chen CN, Jeng SF, Su YN, Chen CY, Chou HC, Tsao PN, Hsieh WS. The sFlt-1/PlGF ratio as a predictor for poor pregnancy and neonatal outcomes. Pediatr Neonatol. 2017 Dec;58(6):529-533. doi: 10.1016/j.pedneo.2016.10.005. Epub 2017 May 10. PMID 28571908
- [Background] Zhao M, Zhu Z, Liu C, Zhang Z. Dual-cutoff of sFlt-1/PlGF ratio in the stratification of preeclampsia: a systematic review and meta-analysis. Arch Gynecol Obstet. 2017 May;295(5):1079-1087. doi: 10.1007/s00404-017-4302-3. Epub 2017 Mar 17. PMID 28314983
- [Background] Stepan H, Herraiz I, Schlembach D, Verlohren S, Brennecke S, Chantraine F, Klein E, Lapaire O, Llurba E, Ramoni A, Vatish M, Wertaschnigg D, Galindo A. Implementation of the sFlt-1/PlGF ratio for prediction and diagnosis of pre-eclampsia in singleton pregnancy: implications for clinical practice. Ultrasound Obstet Gynecol. 2015 Mar;45(3):241-6. doi: 10.1002/uog.14799. No abstract available. PMID 25736847
- [Background] Syngelaki A, Nicolaides KH, Balani J, Hyer S, Akolekar R, Kotecha R, Pastides A, Shehata H. Metformin versus Placebo in Obese Pregnant Women without Diabetes Mellitus. N Engl J Med. 2016 Feb 4;374(5):434-43. doi: 10.1056/NEJMoa1509819. PMID 26840133
- [Background] Rowan JA, Hague WM, Gao W, Battin MR, Moore MP; MiG Trial Investigators. Metformin versus insulin for the treatment of gestational diabetes. N Engl J Med. 2008 May 8;358(19):2003-15. doi: 10.1056/NEJMoa0707193. PMID 18463376
- [Background] Zheng J, Shan PF, Gu W. The efficacy of metformin in pregnant women with polycystic ovary syndrome: a meta-analysis of clinical trials. J Endocrinol Invest. 2013 Nov;36(10):797-802. doi: 10.3275/8932. Epub 2013 Apr 12. PMID 23580001
- [Background] Butalia S, Gutierrez L, Lodha A, Aitken E, Zakariasen A, Donovan L. Short- and long-term outcomes of metformin compared with insulin alone in pregnancy: a systematic review and meta-analysis. Diabet Med. 2017 Jan;34(1):27-36. doi: 10.1111/dme.13150. Epub 2016 Jun 8. PMID 27150509
- [Background] Zhao LP, Sheng XY, Zhou S, Yang T, Ma LY, Zhou Y, Cui YM. Metformin versus insulin for gestational diabetes mellitus: a meta-analysis. Br J Clin Pharmacol. 2015 Nov;80(5):1224-34. doi: 10.1111/bcp.12672. Epub 2015 Jul 14. PMID 25925501
- [Background] Gilbert C, Valois M, Koren G. Pregnancy outcome after first-trimester exposure to metformin: a meta-analysis. Fertil Steril. 2006 Sep;86(3):658-63. doi: 10.1016/j.fertnstert.2006.02.098. Epub 2006 Jul 31. PMID 16879826
- [Background] De Leo V, Musacchio MC, Piomboni P, Di Sabatino A, Morgante G. The administration of metformin during pregnancy reduces polycystic ovary syndrome related gestational complications. Eur J Obstet Gynecol Reprod Biol. 2011 Jul;157(1):63-6. doi: 10.1016/j.ejogrb.2011.03.024. Epub 2011 May 6. PMID 21530058
- [Background] Tan X, Li S, Chang Y, Fang C, Liu H, Zhang X, Wang Y. Effect of metformin treatment during pregnancy on women with PCOS: a systematic review and meta-analysis. Clin Invest Med. 2016 Sep 11;39(4):E120-31. doi: 10.25011/cim.v39i4.27091. PMID 27619399
- [Background] Zhu B, Zhang L, Fan YY, Wang L, Li XG, Liu T, Cao YS, Zhao ZG. Metformin versus insulin in gestational diabetes mellitus: a meta-analysis of randomized clinical trials. Ir J Med Sci. 2016 May;185(2):371-81. doi: 10.1007/s11845-016-1414-x. Epub 2016 Feb 9. PMID 26860118
- [Background] Lautatzis ME, Goulis DG, Vrontakis M. Efficacy and safety of metformin during pregnancy in women with gestational diabetes mellitus or polycystic ovary syndrome: a systematic review. Metabolism. 2013 Nov;62(11):1522-34. doi: 10.1016/j.metabol.2013.06.006. Epub 2013 Jul 23. PMID 23886298
- [Background] Alqudah A, McKinley MC, McNally R, Graham U, Watson CJ, Lyons TJ, McClements L. Risk of pre-eclampsia in women taking metformin: a systematic review and meta-analysis. Diabet Med. 2018 Feb;35(2):160-172. doi: 10.1111/dme.13523. PMID 29044702
- [Background] Chasan-Taber L, Silveira M, Waring ME, Pekow P, Braun B, Manson JE, Solomon CG, Markenson G. Gestational Weight Gain, Body Mass Index, and Risk of Hypertensive Disorders of Pregnancy in a Predominantly Puerto Rican Population. Matern Child Health J. 2016 Sep;20(9):1804-13. doi: 10.1007/s10995-016-1983-3. PMID 27003150
- [Background] Chiswick C, Reynolds RM, Denison F, Drake AJ, Forbes S, Newby DE, Walker BR, Quenby S, Wray S, Weeks A, Lashen H, Rodriguez A, Murray G, Whyte S, Norman JE. Effect of metformin on maternal and fetal outcomes in obese pregnant women (EMPOWaR): a randomised, double-blind, placebo-controlled trial. Lancet Diabetes Endocrinol. 2015 Oct;3(10):778-86. doi: 10.1016/S2213-8587(15)00219-3. Epub 2015 Jul 9. PMID 26165398
- [Background] Dallaglio K, Bruno A, Cantelmo AR, Esposito AI, Ruggiero L, Orecchioni S, Calleri A, Bertolini F, Pfeffer U, Noonan DM, Albini A. Paradoxic effects of metformin on endothelial cells and angiogenesis. Carcinogenesis. 2014 May;35(5):1055-66. doi: 10.1093/carcin/bgu001. Epub 2014 Jan 13. PMID 24419232
- [Background] Zhou G, Myers R, Li Y, Chen Y, Shen X, Fenyk-Melody J, Wu M, Ventre J, Doebber T, Fujii N, Musi N, Hirshman MF, Goodyear LJ, Moller DE. Role of AMP-activated protein kinase in mechanism of metformin action. J Clin Invest. 2001 Oct;108(8):1167-74. doi: 10.1172/JCI13505. PMID 11602624
- [Background] Viollet B, Guigas B, Sanz Garcia N, Leclerc J, Foretz M, Andreelli F. Cellular and molecular mechanisms of metformin: an overview. Clin Sci (Lond). 2012 Mar;122(6):253-70. doi: 10.1042/CS20110386. PMID 22117616
- [Background] Rena G, Hardie DG, Pearson ER. The mechanisms of action of metformin. Diabetologia. 2017 Sep;60(9):1577-1585. doi: 10.1007/s00125-017-4342-z. Epub 2017 Aug 3. PMID 28776086
- [Background] Romero R, Erez O, Huttemann M, Maymon E, Panaitescu B, Conde-Agudelo A, Pacora P, Yoon BH, Grossman LI. Metformin, the aspirin of the 21st century: its role in gestational diabetes mellitus, prevention of preeclampsia and cancer, and the promotion of longevity. Am J Obstet Gynecol. 2017 Sep;217(3):282-302. doi: 10.1016/j.ajog.2017.06.003. Epub 2017 Jun 12. PMID 28619690
- [Background] Chaussabel D, Baldwin N. Democratizing systems immunology with modular transcriptional repertoire analyses. Nat Rev Immunol. 2014 Apr;14(4):271-80. doi: 10.1038/nri3642. PMID 24662387
- [Background] Ribatti D. The discovery of the placental growth factor and its role in angiogenesis: a historical review. Angiogenesis. 2008;11(3):215-21. doi: 10.1007/s10456-008-9114-4. Epub 2008 Jun 21. PMID 18568405
- See also: Maternal, Newborn and Infant Clinical Outcome Review Programme — http://www.hqip.org.uk/national-programmes/

DOCUMENTS (2):
  • Study Protocol and Informed Consent Form (2020-09-07): https://cdn.clinicaltrials.gov/large-docs/13/NCT04855513/Prot_ICF_000.pdf
  • Statistical Analysis Plan (2020-09-07): https://cdn.clinicaltrials.gov/large-docs/13/NCT04855513/SAP_001.pdf